CLINICAL TRIAL: NCT04429945
Title: Immersive Virtual Reality to Improve Outcomes in Patients With Stroke: A Pilot Study
Brief Title: Immersive Virtual Reality in Stroke Pilot Study
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N3449-P; I21RX003449 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: stroke; virtual reality; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Once patients are enrolled, baseline data and pre-intervention outcome measures will be collected. APPs will be selected from the VR Toolkit that best address the individual patient's treatment goals.
  Patients will be instructed in the use of the head mounted display with VR APPs. VR dosage will be two one-half hour sessions per therapy day. Patients can initiate use of a more challenging APPs that gradually includes hand/arm movement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Immersive Virtual Reality (Experimental): A Virtual Reality headset will be used for 30 minutes twice per day outside of usual therapy times while in bed with bedrails raised. Virtual Reality games will be selected that will help with relaxation, pain, and arm and hand recovery after a stroke.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Headset with Virtual Reality Applications
  Other Names: Oculus Quest

SUMMARY:
Over 15,000 Veterans are treated by the VA for stroke each year. A stroke means that part of the brain dies. Many people who have a stroke have difficulty with moving their arm, using their hand, and they have pain. Virtual reality is a video-game based treatment that may help people with stroke improve in these areas. Virtual reality involves using a computer and goggles to make a person feel like they are in a different world with new sights and sounds, relaxing on a beach where there is no pain, or playing the piano. In virtual reality, stroke patients can practice movement in a safe and motivating environment. For example, a person with stroke who has weakness in his/her arm can safely reach for plates in a virtual cupboard. In a virtual environment, the plates can't break. This study will help investigators to determine if people with strokes who are treated with virtual reality like it, and if they have less pain and better movement.

DETAILED DESCRIPTION:
Background. Over the last decade, Virtual Reality (VR) has emerged as a cutting-edge technology in stroke rehabilitation. VR is defined as a type of user-computer interface that implements real-time simulation of an activity or environment allowing user interaction via multiple sensory modalities. VR interventions in a stroke population have been shown to be equivalent to usual care therapies and to enhance motor recovery when utilized as an adjunct. Significance/Impact/Innovation. This research will advance knowledge in rehabilitation research by testing state-of-the-art immersive 3-dimensional VR technology with the post-acute stroke Veteran population. The proposed project addresses: (1) the RR&D goal of maximizing functional recovery, (2) interest in non-pharmacological activity-based interventions for pain, and (3) supports modernization of the Veterans' Health Administration by incorporating technology-assisted rehabilitation.

Specific Aims. (1) Determine the feasibility and tolerability of using a therapeutic VR platform in an inpatient comprehensive stroke rehabilitation program and (2) Estimate the initial clinical efficacy, or effect size, associated with the VR platform using APPS for distraction and upper extremity exercise for Veterans post-stroke.

Methodology. Prospective within-subject pre-post pilot and survey study designs will be used. The target populations are (1) clinical staff who work on the Comprehensive Interdisciplinary Inpatient Rehabilitation Program (CIIRP) at the James A. Haley Veterans' Hospital (JAHVH) in Tampa (sample size N=10) and Veterans who are inpatients in the CIIRP (sample size N=10). The VR intervention consists of wearing a head mounted display that plays APPs ranging from music and nature views for pain distraction to more challenging strengthening and coordination activities such as playing the piano virtually. The intervention will last four weeks. The analytic approach will use descriptive statistics and qualitative methods. Aim 1 will administer a survey with open and closed ended questions to clinicians to examine the feasibility of successfully integrating a VR intervention into the flow of usual care. Feasibility constructs include adaptability (can VR intervention be adapted to an inpatient unit), patient need (do Veterans like and benefit from the intervention), and staff comments/impressions. Responses for each construct will be entered into an excel spreadsheet, one tab for each construct. Responses will then be grouped by similar content. Results will be reported as themes and subthemes. Aim 1 will also track patient VR tolerability by documenting and discussing patient complaints and adverse events. Tolerability data will be extracted from meeting minutes and grouped by similar occurrences. Results will be reported as themes and subthemes. Aim 2 will estimate effect sizes and degree of precision for upper extremity neurologic recovery, hand dexterity, and pain outcomes measured pre and post VR intervention. Neurologic recovery is measured with the Fugl-Meyer Assessment of Motor Recovery after Stroke-Upper Extremity, dexterity is measured with the Action Research Arm Test, and pain is measured with the Pain Outcomes Questionnaire-VA. Because standard scores do not necessarily translate to meaningful clinical differences (improvements), the investigators will identify the proportion of subjects who experience the minimal clinically important difference (MCID). Metrics will also be compared across outcomes.

Next Steps/Implementation. Our next step is to work with our Program Partner in the Physical Medicine and Rehabilitation Office to conduct a large multi-site clinical trial that will incorporate the lessons learned from this feasibility pilot study to test the efficacy of a VR intervention in inpatient rehabilitation and transition to home environments.

ELIGIBILITY:
Inclusion Criteria:

-Veterans who have been diagnosed with

* an acute ischemic or hemorrhagic stroke and
* post-stroke are admitted to James A. Haley Veterans' Hospital inpatient rehabilitation
* age 18-80 with stroke diagnosis verified by brain imaging.

Exclusion Criteria:

* Unable to follow instructions or participate in immersive VR therapy due to significant cognitive impairment,
* History of seizures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna E. Tran, MD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tieri G, Morone G, Paolucci S, Iosa M. Virtual reality in cognitive and motor rehabilitation: facts, fiction and fallacies. Expert Rev Med Devices. 2018 Feb;15(2):107-117. doi: 10.1080/17434440.2018.1425613. Epub 2018 Jan 10. PMID 29313388
- [Background] Lohse KR, Hilderman CG, Cheung KL, Tatla S, Van der Loos HF. Virtual reality therapy for adults post-stroke: a systematic review and meta-analysis exploring virtual environments and commercial games in therapy. PLoS One. 2014 Mar 28;9(3):e93318. doi: 10.1371/journal.pone.0093318. eCollection 2014. PMID 24681826
- [Background] Kiper P, Szczudlik A, Agostini M, Opara J, Nowobilski R, Ventura L, Tonin P, Turolla A. Virtual Reality for Upper Limb Rehabilitation in Subacute and Chronic Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 May;99(5):834-842.e4. doi: 10.1016/j.apmr.2018.01.023. Epub 2018 Feb 14. PMID 29453980
- [Background] Lee MM, Lee KJ, Song CH. Game-Based Virtual Reality Canoe Paddling Training to Improve Postural Balance and Upper Extremity Function: A Preliminary Randomized Controlled Study of 30 Patients with Subacute Stroke. Med Sci Monit. 2018 Apr 27;24:2590-2598. doi: 10.12659/MSM.906451. PMID 29702630
- [Background] Perez-Marcos D, Chevalley O, Schmidlin T, Garipelli G, Serino A, Vuadens P, Tadi T, Blanke O, Millan JDR. Increasing upper limb training intensity in chronic stroke using embodied virtual reality: a pilot study. J Neuroeng Rehabil. 2017 Nov 17;14(1):119. doi: 10.1186/s12984-017-0328-9. PMID 29149855
- [Background] Askin A, Atar E, Kocyigit H, Tosun A. Effects of Kinect-based virtual reality game training on upper extremity motor recovery in chronic stroke. Somatosens Mot Res. 2018 Mar;35(1):25-32. doi: 10.1080/08990220.2018.1444599. Epub 2018 Mar 13. PMID 29529919
- [Background] Paquin K, Crawley J, Harris JE, Horton S. Survivors of chronic stroke - participant evaluations of commercial gaming for rehabilitation. Disabil Rehabil. 2016 Oct;38(21):2144-52. doi: 10.3109/09638288.2015.1114155. Epub 2016 Jan 5. PMID 26728133
- [Background] Kong KH, Loh YJ, Thia E, Chai A, Ng CY, Soh YM, Toh S, Tjan SY. Efficacy of a Virtual Reality Commercial Gaming Device in Upper Limb Recovery after Stroke: A Randomized, Controlled Study. Top Stroke Rehabil. 2016 Oct;23(5):333-40. doi: 10.1080/10749357.2016.1139796. Epub 2016 Apr 21. PMID 27098818
- [Background] Lai SM, Studenski S, Duncan PW, Perera S. Persisting consequences of stroke measured by the Stroke Impact Scale. Stroke. 2002 Jul;33(7):1840-4. doi: 10.1161/01.str.0000019289.15440.f2. PMID 12105363
- [Background] Saposnik G, Cohen LG, Mamdani M, Pooyania S, Ploughman M, Cheung D, Shaw J, Hall J, Nord P, Dukelow S, Nilanont Y, De Los Rios F, Olmos L, Levin M, Teasell R, Cohen A, Thorpe K, Laupacis A, Bayley M; Stroke Outcomes Research Canada. Efficacy and safety of non-immersive virtual reality exercising in stroke rehabilitation (EVREST): a randomised, multicentre, single-blind, controlled trial. Lancet Neurol. 2016 Sep;15(10):1019-27. doi: 10.1016/S1474-4422(16)30121-1. Epub 2016 Jun 27. PMID 27365261
- [Background] Saposnik G, Levin M; Outcome Research Canada (SORCan) Working Group. Virtual reality in stroke rehabilitation: a meta-analysis and implications for clinicians. Stroke. 2011 May;42(5):1380-6. doi: 10.1161/STROKEAHA.110.605451. Epub 2011 Apr 7. PMID 21474804
- [Background] Palma GC, Freitas TB, Bonuzzi GM, Soares MA, Leite PH, Mazzini NA, Almeida MR, Pompeu JE, Torriani-Pasin C. Effects of virtual reality for stroke individuals based on the International Classification of Functioning and Health: a systematic review. Top Stroke Rehabil. 2017 May;24(4):269-278. doi: 10.1080/10749357.2016.1250373. Epub 2016 Oct 31. PMID 27796177
- [Background] Glegg SMN, Levac DE. Barriers, Facilitators and Interventions to Support Virtual Reality Implementation in Rehabilitation: A Scoping Review. PM R. 2018 Nov;10(11):1237-1251.e1. doi: 10.1016/j.pmrj.2018.07.004. PMID 30503231
- [Background] Yates M, Kelemen A, Sik Lanyi C. Virtual reality gaming in the rehabilitation of the upper extremities post-stroke. Brain Inj. 2016;30(7):855-63. doi: 10.3109/02699052.2016.1144146. Epub 2016 Mar 30. PMID 27029647
- [Background] Ikbali Afsar S, Mirzayev I, Umit Yemisci O, Cosar Saracgil SN. Virtual Reality in Upper Extremity Rehabilitation of Stroke Patients: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2018 Dec;27(12):3473-3478. doi: 10.1016/j.jstrokecerebrovasdis.2018.08.007. Epub 2018 Sep 5. PMID 30193810
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Aminov A, Rogers JM, Middleton S, Caeyenberghs K, Wilson PH. What do randomized controlled trials say about virtual rehabilitation in stroke? A systematic literature review and meta-analysis of upper-limb and cognitive outcomes. J Neuroeng Rehabil. 2018 Mar 27;15(1):29. doi: 10.1186/s12984-018-0370-2. PMID 29587853
- [Background] Choi YH, Ku J, Lim H, Kim YH, Paik NJ. Mobile game-based virtual reality rehabilitation program for upper limb dysfunction after ischemic stroke. Restor Neurol Neurosci. 2016 May 2;34(3):455-63. doi: 10.3233/RNN-150626. PMID 27163250
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Paolucci S, Iosa M, Toni D, Barbanti P, Bovi P, Cavallini A, Candeloro E, Mancini A, Mancuso M, Monaco S, Pieroni A, Recchia S, Sessa M, Strambo D, Tinazzi M, Cruccu G, Truini A; Neuropathic pain special interest group of the Italian Neurological Society. Prevalence and Time Course of Post-Stroke Pain: A Multicenter Prospective Hospital-Based Study. Pain Med. 2016 May;17(5):924-30. doi: 10.1093/pm/pnv019. Epub 2015 Dec 14. PMID 26814255
- [Background] Malfliet A, Coppieters I, Van Wilgen P, Kregel J, De Pauw R, Dolphens M, Ickmans K. Brain changes associated with cognitive and emotional factors in chronic pain: A systematic review. Eur J Pain. 2017 May;21(5):769-786. doi: 10.1002/ejp.1003. Epub 2017 Feb 1. PMID 28146315
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Jin W, Choo A, Gromala D, Shaw C, Squire P. A Virtual Reality Game for Chronic Pain Management: A Randomized, Controlled Clinical Study. Stud Health Technol Inform. 2016;220:154-60. PMID 27046570
- [Background] Gold JI, Belmont KA, Thomas DA. The neurobiology of virtual reality pain attenuation. Cyberpsychol Behav. 2007 Aug;10(4):536-44. doi: 10.1089/cpb.2007.9993. PMID 17711362
- [Background] Garrett B, Taverner T, Gromala D, Tao G, Cordingley E, Sun C. Virtual Reality Clinical Research: Promises and Challenges. JMIR Serious Games. 2018 Oct 17;6(4):e10839. doi: 10.2196/10839. PMID 30333096
- [Background] Garrett B, Taverner T, Masinde W, Gromala D, Shaw C, Negraeff M. A rapid evidence assessment of immersive virtual reality as an adjunct therapy in acute pain management in clinical practice. Clin J Pain. 2014 Dec;30(12):1089-98. doi: 10.1097/AJP.0000000000000064. PMID 24535053
- [Background] Kleim JA, Jones TA. Principles of experience-dependent neural plasticity: implications for rehabilitation after brain damage. J Speech Lang Hear Res. 2008 Feb;51(1):S225-39. doi: 10.1044/1092-4388(2008/018). PMID 18230848
- [Background] Arya KN, Pandian S, Verma R, Garg RK. Movement therapy induced neural reorganization and motor recovery in stroke: a review. J Bodyw Mov Ther. 2011 Oct;15(4):528-37. doi: 10.1016/j.jbmt.2011.01.023. Epub 2011 Feb 25. PMID 21943628
- [Background] Sunderland A, Tinson DJ, Bradley EL, Fletcher D, Langton Hewer R, Wade DT. Enhanced physical therapy improves recovery of arm function after stroke. A randomised controlled trial. J Neurol Neurosurg Psychiatry. 1992 Jul;55(7):530-5. doi: 10.1136/jnnp.55.7.530. PMID 1640226
- [Background] Garrett B, Taverner T, McDade P. Virtual Reality as an Adjunct Home Therapy in Chronic Pain Management: An Exploratory Study. JMIR Med Inform. 2017 May 11;5(2):e11. doi: 10.2196/medinform.7271. PMID 28495661
- [Background] Duncan P, Studenski S, Richards L, Gollub S, Lai SM, Reker D, Perera S, Yates J, Koch V, Rigler S, Johnson D. Randomized clinical trial of therapeutic exercise in subacute stroke. Stroke. 2003 Sep;34(9):2173-80. doi: 10.1161/01.STR.0000083699.95351.F2. Epub 2003 Aug 14. PMID 12920254
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] Hylin MJ, Kerr AL, Holden R. Understanding the Mechanisms of Recovery and/or Compensation following Injury. Neural Plast. 2017;2017:7125057. doi: 10.1155/2017/7125057. Epub 2017 Apr 20. PMID 28512585
- [Background] Dimyan MA, Cohen LG. Neuroplasticity in the context of motor rehabilitation after stroke. Nat Rev Neurol. 2011 Feb;7(2):76-85. doi: 10.1038/nrneurol.2010.200. Epub 2011 Jan 18. PMID 21243015
- [Background] Merians AS, Jack D, Boian R, Tremaine M, Burdea GC, Adamovich SV, Recce M, Poizner H. Virtual reality-augmented rehabilitation for patients following stroke. Phys Ther. 2002 Sep;82(9):898-915. PMID 12201804
- [Background] Birckhead B, Khalil C, Liu X, Conovitz S, Rizzo A, Danovitch I, Bullock K, Spiegel B. Recommendations for Methodology of Virtual Reality Clinical Trials in Health Care by an International Working Group: Iterative Study. JMIR Ment Health. 2019 Jan 31;6(1):e11973. doi: 10.2196/11973. PMID 30702436
- [Background] Fodor LA, Cotet CD, Cuijpers P, Szamoskozi S, David D, Cristea IA. The effectiveness of virtual reality based interventions for symptoms of anxiety and depression: A meta-analysis. Sci Rep. 2018 Jul 9;8(1):10323. doi: 10.1038/s41598-018-28113-6. PMID 29985400
- [Background] Kwakkel G, van Peppen R, Wagenaar RC, Wood Dauphinee S, Richards C, Ashburn A, Miller K, Lincoln N, Partridge C, Wellwood I, Langhorne P. Effects of augmented exercise therapy time after stroke: a meta-analysis. Stroke. 2004 Nov;35(11):2529-39. doi: 10.1161/01.STR.0000143153.76460.7d. Epub 2004 Oct 7. PMID 15472114
- [Background] Fowler CA, Ballistrea LM, Mazzone KE, Martin AM, Kaplan H, Kip KE, Murphy JL, Winkler SL. A virtual reality intervention for fear of movement for Veterans with chronic pain: protocol for a feasibility study. Pilot Feasibility Stud. 2019 Dec 11;5:146. doi: 10.1186/s40814-019-0501-y. eCollection 2019. PMID 31890259
- [Background] Fowler CA, Ballistrea LM, Mazzone KE, Martin AM, Kaplan H, Kip KE, Ralston K, Murphy JL, Winkler SL. Virtual Reality as a Therapy Adjunct for Fear of Movement in Veterans With Chronic Pain: Single-Arm Feasibility Study. JMIR Form Res. 2019 Oct 30;3(4):e11266. doi: 10.2196/11266. PMID 31670696
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Lang CE, Edwards DF, Birkenmeier RL, Dromerick AW. Estimating minimal clinically important differences of upper-extremity measures early after stroke. Arch Phys Med Rehabil. 2008 Sep;89(9):1693-700. doi: 10.1016/j.apmr.2008.02.022. PMID 18760153
- [Background] Simpson LA, Eng JJ. Functional recovery following stroke: capturing changes in upper-extremity function. Neurorehabil Neural Repair. 2013 Mar-Apr;27(3):240-50. doi: 10.1177/1545968312461719. Epub 2012 Oct 16. PMID 23077144
- [Background] Page SJ, Fulk GD, Boyne P. Clinically important differences for the upper-extremity Fugl-Meyer Scale in people with minimal to moderate impairment due to chronic stroke. Phys Ther. 2012 Jun;92(6):791-8. doi: 10.2522/ptj.20110009. Epub 2012 Jan 26. PMID 22282773
- [Background] Clark ME, Gironda RJ, Young RW. Development and validation of the Pain Outcomes Questionnaire-VA. J Rehabil Res Dev. 2003 Sep-Oct;40(5):381-95. doi: 10.1682/jrrd.2003.09.0381. PMID 15080223
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Morris SB, DeShon RP. Combining effect size estimates in meta-analysis with repeated measures and independent-groups designs. Psychol Methods. 2002 Mar;7(1):105-25. doi: 10.1037/1082-989x.7.1.105. PMID 11928886
- [Background] Barak S, Duncan PW. Issues in selecting outcome measures to assess functional recovery after stroke. NeuroRx. 2006 Oct;3(4):505-24. doi: 10.1016/j.nurx.2006.07.009. PMID 17012065
- See also: SAS Macro for Effects Size Computations — https://analytics.ncsu.edu/sesug/2012/SD-06.pdf
- See also: Market projections for VR in Healthcare — https://www.reportsanddata.com/report-detail/virtual-reality-in-healthcare-market

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans diagnosed with an acute ischemic or hemorrhagic stroke who were admitted to James A. Haley VA Hospital inpatient rehabilitation were recruited from 6/17/21 thru 9/7/22. Potential subjects were identified by the Physical Medicine & Rehabilitation Physician, PI Tran, or the study coordinator in Dr. Tran's absence. The PI and/or study coordinator used a HIPAA Waiver and a Waiver of Informed Consent to review inclusion/exclusion criteria with the medical records to determine eligibility.
Pre-assignment Details: No participants were excluded from study participation. This was due to inclusion/exclusion criteria alignment with admission criteria for the inpatient stroke rehabilitation program. The post-treatment measurement period was reduced from week 4 to week 3 secondary to COVID-19 hospital policies which prioritized shorter inpatient stays when feasible. Specifically, the hospital triage approach prioritized inpatient beds for COVID-19 patients
Groups:
- Single Arm Within-participants Pre-post: The VR intervention uses off the shelf technology: Oculus Quest Head Mounted Display and commercially available APPs specifically developed or adapted for Oculus Quest. APP selection for individual patients will be guided by motor difficulty of the APPs. As tolerated, patients will advance to more difficult APPs which require hand and finger movement, with the high-level APPs requiring controlled movement. Participants will be measures at inpatient stroke rehabilitation program entry (baseline) and and again upon program discharge (post).
Period: Overall Study
Arm/Group | Single Arm Within-participants Pre-post
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The target population was Veterans receiving care for a stroke in a Comprehensive Interdisciplinary Inpatient Rehabilitation Program.
Arm/Group | Single Arm Within-participants Pre-post
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Fugl-Meyer Assessment of Motor Recovery after Stroke-Upper Extremity [Mean (Standard Deviation); unit: Units on a Scale] — The 63-item Fugl-Meyer Assessment of Motor Recovery after Stroke-Upper Extremity is a measure of upper extremity stroke recovery, specifically functional impairment across 4 sub-domains: Joint Pain, Motor Function, Passive Joint Range of Motion, and Sensation. Each functional test is rated on a 0 to 2 scale with higher scores indicating greater function. Test scores were summed within each sub-domain: Joint Pain = 0-24, Motor Function = 0-66; Passive Joint Range of Motion = 0-24; Sensation = 0-12. Within each sub-domain, higher scores indicate greater improvement in upper extremity function.
  Units on a Scale
    Joint Pain | 21.40 (3.53)
    Motor Function | 45.70 (20.95)
    Passive Joint ROM | 22.80 (2.70)
    Sensation | 11.20 (1.69)
Action Research Arm Test [Mean (Standard Deviation); unit: Units on a Scale] — The Action Research Arm Test includes 19 tests across 4 sub-domains: Grasp, Grip, Pinch, Gross Movement. Each test is scored on a 0 (no movement possible) to 3 (movement performed normally) scale. Within each domain a score of 3 on the first and hardest test, the remaining tests are also scored as 3. A score of 0 on the second, easiest test, remaining tests are scored as 0. Tests are summed for each domain: Grasp= 0-18, Grip= 0-12; Pinch= 0-18; Gross Movement= 0-9. A total score is then summed from sub-domains (range= 0-57) with higher scores indicating better hand dexterity.
  Units on a Scale | 29.60 (22.68)
Pain Outcomes Questionnaire for Veterans - Pain Numeric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The 0 (no pain at all) to 10 (worst pain possible) pain numeric rating scale from the Pain Outcomes Questionnaire-VA was used to measure post-stroke pain intensity.
  units on a scale | 1.40 (2.67)

OUTCOME MEASURES:

1. Primary Outcome: Action Research Arm Test
Description: The Action Research Arm Test includes 19 clinician-administered tests across 4 sub-domains: Grasp, Grip, Pinch, Gross Movement. Each test is scored on a 0 (no movement possible) to 3 (movement performed normally) scale. Within each domain a score of 3 on the first and hardest test, the remaining tests are also scored as 3. A score of 0 on the second, easiest test, remaining tests are scored as 0. Tests are summed within each domain: Grasp (range = 0-18), Grip (range = 0-12); Pinch (range = 0-18); Gross Movement (range = 0-9). A total score was then calculated by summing the scores from each sub-domains (range= 0-57) with higher scores indicating better hand dexterity.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Single Arm Within-participants Pre-post
Number analyzed (Participants) | 10
Units on a Scale | 38.80 (22.03)

2. Primary Outcome: Fugl-Meyer Assessment Upper Extremity
Description: The Fugl-Meyer Assessment of Motor Recovery after Stroke-Upper Extremity is a measure of upper extremity stroke recovery, specifically functional impairment. It consists of 63 functional rests across 4 sub-domains: Joint Pain, Motor Function, Passive Joint Range of Motion, and Sensation. Each functional test is rated on a 0 to 2 scale with higher scores indicating greater functioning. Test scores were then summed within each sub-domain: Joint Pain (range = 0-24), Motor Function (range = 0-66); Passive Joint Range of Motion (range = 0-24); Sensation (range = 0-12). Within each sub-domain, higher scores indicate greater improvement in upper extremity function.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Single Arm Within-participants Pre-post
Number analyzed (Participants) | 10
Units on a Scale
  Joint Pain | 21.60 (3.63)
  Motor Function | 51.90 (18.64)
  Passive Joint ROM | 23.20 (1.69)
  Sensation | 11.60 (0.84)

3. Secondary Outcome: Pain Outcomes Questionnaire-VA
Description: The 0 (no pain at all) to 10 (worst pain possible) pain numeric rating scale from the Pain Outcomes Questionnaire-VA was used to measure post-stroke pain intensity.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Within-participants Pre-post
Number analyzed (Participants) | 10
units on a scale | 0.90 (2.23)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected across the entire study, up to 15 months.
Description: The therapeutic risks to subjects include the potential for "cybersickness" (e.g. vertigo, nausea), emotional adverse effects (e.g. fear, anxiety) and discomfort or inconvenience related to the VR equipment (e.g. ill-fitting headset, facial pain). VR, in general, is well tolerated and risks to subjects are expected to be small and, if present, mild in severity. The advantage of implementing this intervention in an inpatient environment is that adverse events can be immediately addressed.
Groups:
- Single Arm Within-participants Pre-post: The VR intervention uses off the shelf technology: Oculus Quest Head Mounted Display and commercially available APPs specifically developed or adapted for Oculus Quest. APP selection for individual patients will be guided by motor difficulty of the APPs. As tolerated, patients will advance to more difficult APPs which require hand and finger movement, with the high-level APPs requiring controlled movement. Participants will be measured at inpatient stroke rehabilitation program entry (baseline) and and again upon program discharge (post).
Arm/Group | Single Arm Within-participants Pre-post
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Within-participants Pre-post (N=10)
Cybersickness (Ear and labyrinth disorders) | 1 (2) — Virtual reality induced dizziness, nausea, or motion sickness.
Headset discomfort. (Product Issues) | 1 (4) — Discomfort or inconvenience related to the VR equipment (e.g. ill-fitting headset, facial pain). Subject felt itchiness on bridge of nose. Research staff placed band-aid on the bridge of participants nose to prevent itchiness.

LIMITATIONS AND CAVEATS:
COVID-19 hospital policy contributed to slow recruitment, reduced inpatient stays, and competition for beds. Low referral rates led to more higher functioning patients. Unreliable hospital Wifi presented challenges for using VR APPs and installing updates. Team competed for treatment times with clinical staff. Thus, twice daily sessions were often completed back-to-back. Storing devices in locked offices per IRB protocol limited clinical staff access to technology for further use with Veterans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04429945/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04429945/ICF_000.pdf